CLINICAL TRIAL: NCT01899716
Title: Exercise and Severe Depression: Clinical and Biological Analysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07-438
Record Dates: First submitted 2013-06-13; First posted 2013-07-15 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-05

CONDITIONS: Depression
Keywords: Severe Depression; Quality of life; Exercise; BDNF; TBARS
MeSH Terms: conditions — Depression; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Exercise (Experimental): Aerobic Exercise, 3 times peer week, A dose of 16.5 kcal/kg weight peer week.
  Interventions: Other: Exercise
- Control (No Intervention)

INTERVENTIONS:
Other: Exercise
  Other Names: Aerobic Exercise
  Arms: Exercise

SUMMARY:
The study aimed to evaluate the use of exercise as a complementary strategy to treat severe major depression in inpatients.

Hypothesis: Exercise can be used as a safe and efficacious complimentary strategy in severe depressed inpatients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Major Depressive Disorder according to M.I.N.I (DSM-IV) criteria American Psychiatry Association(1994)
* score of 25 or more on Hamilton-17
* not being involved in other physical activity programs during the hospitalization
* aged between 18 and 60 years
* being able to read, understand, and provide written informed consent

Exclusion Criteria:

* have three or more cardiovascular risk factors according to Physical Activity Readiness Questionnaire (PAR-Q)
* are unable to exercise due other clinical condition
* have diagnosis of Schizophrenia, Bipolar disorder or current use of alcohol or other drugs according to M.I.N.I DSM-IV criteria American Psychiatry Association(1994)
* if they are taking beta-blocking medications

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2008-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms | 2 weeks of hospitalization (14 days)
  Hamilton 17 for depression

SECONDARY OUTCOMES:
Quality of Life | Baseline, after 2 weeks of hospitalization and at discharge (participants will be followed for the duration of hospital stay, an expected average of 3 weeks)
  WHOQOL-BREF
Brain-Derived Neurotrophic Factor(BDNF) | Baseline, after 2 weeks of hospitalization and at discharge (participants will be followed for the duration of hospital stay, an expected average of 3 weeks)
Thiobarbituric acid reactive substances(TBARS) | Baseline, after 2 weeks of hospitalization and at discharge (participants will be followed for the duration of hospital stay, an expected average of 3 weeks)
Depressive symptoms at discharge (participants will be followed for the duration of hospital stay, an expected average of 3 weeks) | Discharge
  Hamilton Scores at discharge

CONTACTS AND LOCATIONS:
Overall Officials: Felipe B Schuch, MSc, Principal Investigator — HCPA; Marcelo PA Fleck, PhD, Study Director — HCPA
Locations (1):
- Hospital de Clincas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Result] Schuch FB, Vasconcelos-Moreno MP, Borowsky C, Fleck MP. Exercise and severe depression: preliminary results of an add-on study. J Affect Disord. 2011 Oct;133(3):615-8. doi: 10.1016/j.jad.2011.04.030. Epub 2011 May 25. PMID 21616540
- [Result] Schuch FB, de Almeida Fleck MP. Is Exercise an Efficacious Treatment for Depression? A Comment upon Recent Negative Findings. Front Psychiatry. 2013 Apr 2;4:20. doi: 10.3389/fpsyt.2013.00020. eCollection 2013. No abstract available. PMID 23565097